CLINICAL TRIAL: NCT00587353
Title: Tobacco Use Intervention Among Radiation Oncology Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Yolanda I. Garces, MD, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-006180
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Tobacco Use Disorder
Keywords: tobacco use cessation; radiation oncology; smoking
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Behavioral and pharmacologic tobacco use intervention — A novel approach to providing an intervention for tobacco users who are receiving radiation therapy is to provide an individual tobacco use intervention that utilizes concepts of motivational interviewing strategies to facilitate self-exploration of the reasons for continued smoking and a treatment plan that is comprehensive and builds self-efficacy, provides one-on-one counseling, and includes tobacco treatment pharmacotherapies. The pharmacotherapies will be tailored to the patients needs. One could utilize varenicline, bupropion, and/or nicotine replacement therapies.

SUMMARY:
Tobacco prevention and intervention strategies in the general population are ongoing and evolving. However, strategies to help cancer patients overcome tobacco dependence have been limited. Radiation oncology patients who continue to smoke despite their cancer diagnosis have a lower quality of life (QOL), increased frequency and severity of side effects during their cancer treatment, higher risks of developing a smoking-related primary cancer, and may have a poorer survival rate than their non-smoking counterparts. These are all compelling reasons to be more pro-active in helping cancer patients stop smoking. The overall objective of this project is to adapt a model of an effective tobacco use intervention that can be delivered by any trained radiation oncologist and their staff.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age;
* current cigarette smoker (smoked any cigarettes within the previous 7 days prior to their first visit) or recent ex-smoker (last cigarette smoked was >7 but ≤ 30 days);
* planning to undergo radiation therapy (RT) that is to be delivered by the members of the Department of Radiation Oncology in Rochester, MN;
* be receiving a minimum of 5 weeks of RT and/or be willing to return for all 5 sessions.

Exclusion Criteria:

* patient is currently (in previous 30 days) using other formal behavioral tobacco cessation program [i.e., behavioral therapy (Nicotine Dependence Consultation and treatment) or telephone quitline];
* daily use of tobacco products other than cigarettes;
* hospitalized patients;
* Karnofsky Performance Status (KPS) score of < 60 (KPS = 60 corresponds to a person who requires occasional assistance but is able to care for most of their own needs;
* presence of an unstable or untreated psychiatric disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary aim is to pilot test the intervention in radiation oncology patients (N=30). The primary dependent measure is self-reported 7-day point prevalence tobacco abstinence confirmed with expired air carbon monoxide. | 6 months

SECONDARY OUTCOMES:
We will be collecting data on QOL and psychosocial measures. This data will be reported descriptively and will be collected on our future study with appropriate statistical analyses. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda I Garces, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States